CLINICAL TRIAL: NCT01626261
Title: Study of Provocation Concerning Implants´Safety in Electronic and Magnetic Fields in Their Environment
Brief Title: Examination of Implant´s Safety in an Electronic and Magnetic Field Environment
Acronym: FEMU
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 09-051
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Disorder of Cardiac Pacemaker System; Disorder of Implantable Defibrillator; Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood (serum and plasma) urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac pacemaker
  Interventions: Device: Magnetic and electric field´s impact on the implant

INTERVENTIONS:
Device: Magnetic and electric field´s impact on the implant — Examination of magnetic and electric field's impact on the implant regarding: stability detection threshold using different strength of magnetic and electric field
  Other Names: Examination

SUMMARY:
The number of active electrical cardiac implants such as internal cardioverter defibrillators (ICDs), pacemakers or cardiac contractility modules (CCM) has significantly risen over the last two decades. This has been paralleled by an increase in the number of sources of electromagnetic fields in daily life and occupational circumstances.

To date it remains unclear whether patients are at risk of device failure when being subjected to these fields. There are currently no general guidelines available to help clinicians informing their patients about safety levels and behavior around these electromagnetic fields.

This study aims to identify the thresholds of safe use of these devices and potential failures under worst-case conditions in 50/60 Hz fields (i.e.

power line frequency). Device implanted patients will be exposed to electric, magnetic and combined fields of different intensity at various device programming (e.g. nominal and maximum sensitivity). The results will show whether patients are safe in public or occupational environments, which medical relevant disturbances can occur and if a correlation exists between disturbances and device type or patients physique.

ELIGIBILITY:
Inclusion Criteria:

* men and women between 18 and 80 years
* Implantation of a Pacemaker (SM)-/ ICD-assembly at least four weeks ago
* signed informed consent

Exclusion Criteria:

* enduring addiction of implant
* thyroid disease
* electrolyte imbalance on the trial day
* pregnancy and breastfeeding
* acute myocardial infarction (<30 days)
* Comorbidity, which complicates an emergency assistance, e.g. morbus bechterew, glaucoma, micturition disturbance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age between 18 and 80
Sampling Method: Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2009-09; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Interference threshold of the device in electromagnetic fields in V/m and/or µT | for every patient during one ambulant visit about 1 hour study examination

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Napp, MD, Principal Investigator — University Hospital, Aachen
Locations (1):
- Universtiy Hospital RWTH Aachen, Aachen, Northrhine-Westfalia, Germany

REFERENCES:
- [Derived] Napp A, Joosten S, Stunder D, Knackstedt C, Zink M, Bellmann B, Marx N, Schauerte P, Silny J. Electromagnetic interference with implantable cardioverter-defibrillators at power frequency: an in vivo study. Circulation. 2014 Jan 28;129(4):441-50. doi: 10.1161/CIRCULATIONAHA.113.003081. Epub 2013 Oct 25. PMID 24163067